CLINICAL TRIAL: NCT03300453
Title: Protocol AMT110-CD-001: A Phase I/II, Open-label, Study of Intracerebral Administration of Adeno-associated Viral Vector Containing the Human Alpha-N-acetylglucosaminidase cDNA in Children With Sanfilippo Type B Syndrome
Brief Title: Intracerebral Gene Therapy in Children With Sanfilippo Type B Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UniQure Biopharma B.V. (Industry)
Collaborators: Venn Life Sciences (Other); Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT110-CD-001
Record Dates: First submitted 2016-06-15; First posted 2017-10-03 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-10

CONDITIONS: Sanfilippo Syndrome B
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rAAV2/5-hNAGLU (Experimental): Each patient will receive 960 µL of vector suspension. The vector suspension will be deposited simultaneously at 16 sites, each deposit containing 2.4x 1011 vg (4x1012 vg in total).
  Interventions: Drug: rAAV2/5-hNAGLU

INTERVENTIONS:
Drug: rAAV2/5-hNAGLU — one-time brain intraparenchymal gene therapy dose
  Other Names: AAV5

SUMMARY:
This is an open-label, phase I/II study of intra-cerebral administration of adenovirus-associated viral vector containing the human NAGLU cDNA to children suffering from Sanfilippo type B syndrome.

DETAILED DESCRIPTION:
This is an open-label, phase I/II study of intra-cerebral administration of adenovirus-associated viral vector containing the human NAGLU cDNA to children suffering from Sanfilippo type B syndrome.

Four patients, 18 months up to the 5th birthday, have been included.

The inclusion period will be 8 to 12 months. The duration of follow-up for each patient is 1 year post-surgery. The duration of the first extension phase is 18 months. The duration of the second extension phase is 36 months. Therefore, the maximum time of the follow-up will be 66 months

ELIGIBILITY:
Inclusion criteria:

* Age: 18 months up to 60 months (5th birthday);
* Onset of clinical manifestations related to mucopolysaccharidosis type IIIB (MPSIIIB);
* NAGLU activity in peripheral blood cell and/or cultured fibroblast extracts of less than 10% of controls;
* Patient affiliated to, or covered by a French social security regimen, or European patients with European Health Insurance Card;
* Family understanding the procedure and the informed consent;
* Signed informed consent by both parents or legal representative;
* Vital laboratory parameters within normal range.

Exclusion Criteria:

* Presence of brain atrophy on baseline MRI judged on a cortico-dural distance of more than 0.6 cm;
* Any condition that would contraindicate general anesthesia;
* Any other permanent medical condition not related to MPSIIIB that could contraindicate the study participation;
* No independent walking (ability to walk without help);
* Any medication aiming at modifying the natural course of MPSIIIB given during the 6 months before vector injection (sleep and mood regulators are accepted);
* Any condition that would contraindicate treatment with Modigraf®, Cellcept® and prednisolone (Solupred® and Solumedrol®).

Ages: 18 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2013-09-17 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related (Serious) Adverse Events as assessed by continuous evaluation of change from baseline | Baseline until end of study (Month 66)
  Multiple measurements will be aggregated to derive the number of participants with Abnormal Laboratory Values and/or Adverse Events that are related to Treatment.

SECONDARY OUTCOMES:
Number of Participants with presence of brain atrophy, white matter lesions and other lesions as assessed by cerebral MRI | Baseline until end of study (Month 66)
  MRIs at Baseline, Month 3, Month 12, Month 30, Month 48 and last visit Month 66.
  Cerebral MRI will be collected for safety assessment to retrospectively evaluate for efficacy at Baseline, D0, Month 3, Month12, Month 30 and last visit Month 66.

CONTACTS AND LOCATIONS:
Overall Officials: Kumaran Deiva, MD, Principal Investigator — Hopitaux Universitaires Paris-Sud
Locations (1):
- Hopitaux Universitaires Paris-Sud, Paris, Le Kremlin-Bicetre Cedex, France

REFERENCES:
- [Derived] Gougeon ML, Poirier-Beaudouin B, Ausseil J, Zerah M, Artaud C, Heard JM, Deiva K, Tardieu M. Cell-Mediated Immunity to NAGLU Transgene Following Intracerebral Gene Therapy in Children With Mucopolysaccharidosis Type IIIB Syndrome. Front Immunol. 2021 May 10;12:655478. doi: 10.3389/fimmu.2021.655478. eCollection 2021. PMID 34040605